CLINICAL TRIAL: NCT02910011
Title: A Phase 2, Exploratory Study to Investigate Safety and Efficacy of Doxycycline Monohydrate Hydrogel (NANODOX® HYDROGEL 1%) In Atopic Dermatitis
Brief Title: Topical NanoDox® for Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Alchem Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601657 - A
Record Dates: First submitted 2016-09-01; First posted 2016-09-21 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Topical Administration of Study Drug (Experimental): 2.5 grams of Nanodox 1% (doxycycline monohydrate hydrogel) will be applied topically to an indicated lesion daily for 28 days
  Interventions: Drug: Nanodox 1% (doxycycline monohydrate hydrogel)

INTERVENTIONS:
Drug: Nanodox 1% (doxycycline monohydrate hydrogel) — Subjects will be asked to apply NanoDOX® Hydrogel 1% once daily at bedtime for up to four weeks or until complete clearance whichever is sooner

SUMMARY:
This study will investigate the safety and clinical efficacy of a novel doxycycline topical formulation in subjects with Atopic Dermatitis (AD). The investigators hypothesize that daily application of the study drug in AD subjects will reduce severity of the disease, by reducing skin driven inflammation and restoring skin barrier function. The investigators will also monitor the anti-microbial activity of this product on AD skin, as colonization with Staph aureus is typically associated with disease severity.

DETAILED DESCRIPTION:
Atopic Dermatitis (AD) is the most common inflammatory skin disease, affecting about 17% of children and 6% adults in the USA , . AD is characterized by skin barrier disruption, an aberrant adaptive immune response (i.e., Th2 polarized) to environmental allergens, susceptibility to cutaneous bacterial infections and intractable itch , . The intense pruritus and cutaneous infections contribute to the morbidity of AD and are major drivers of the reduced quality-of-life associated with this disease , . In the World Health Organization 2010 Global Burden of Disease survey, AD has ranked first among common skin diseases . So far, AD treatments have targeted inflammation with the widespread use of topical and more intermittent use of systemic corticosteroids. In summary, despite its high prevalence, effects on quality-of-life and economic burden - there are few effective treatments for AD.

Doxycycline are tetracycline antibiotics broadly used systemically to treat inflammatory-dermatologic conditions. Several studies in human and animal models have shown doxycycline have anti-inflammatory and pro-healing properties, mainly by blocking tissue proteolytic activity. Doxycycline have been reported to nonselectively inhibit members of the metalloproteinases (MMP) superfamily [reviewed in , ]. In addition to this direct inhibitory activity, doxycycline indirectly prevents tryptic kallikreins activation by MMPs . Growing body of evidence suggests that the tetracycline might also directly downregulate Protease Activator receptor (PAR)-2 expression and function, which was also found to play a role in induction of local inflammatory mediators . Importantly, the doxycycline antimicrobial activity could lead to reduced Staphylococcus infection/colonization in AD skin, a known trigger of AD flares

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 through 65 years of age, inclusive who are generally healthy except for active atopic dermatitis diagnosed by the following criteria.
* Active Atopic Dermatitis: Subjects must have within the last 3 months according to medical records, patient account or by medical exam of the investigator:

  * Pruritus
  * Eczema (acute, subacute, chronic)
  * Chronic or relapsing history

Most subjects will have (seen in most cases, adding support to the diagnosis):

* Early age at onset
* Atopy
* Personal and/or family history
* Xerosis

Subjects may have (these clinical associations help to suggest the diagnosis of AD but are too nonspecific for defining or detecting AD for research or epidemiological studies):

1. Atypical vascular responses (e.g., facial pallor, white dermographism, delayed blanch response)
2. Keratosis pilaris/hyperlinear palms/ichthyosis
3. Ocular/periorbital changes
4. Other regional findings (e.g., perioral changes/periauricular lesions)
5. Perifollicular accentuation/lichenification/prurigo lesions

   * Moderate to Severe AD: clinical score based on Eczema Area and Severity Score (EASI) ≥ 10
   * If receiving antihistamines, are on a stabilized dose, and expect to maintain this dose throughout the study
   * All female subjects of childbearing potential must have a negative pregnancy test at screening visit and must be on an acceptable methods of contraception from the Screening Visit continuously until 30 days after stopping study drug.

Exclusion Criteria:

* As determined by the study doctor, a medical history that may interfere with study objectives (cancer, chronic illness)
* Known allergy to tetracycline
* Subjects with a systemic infection requiring a course of systemic antibiotics or antivirals within the last 2 weeks
* Unstable AD or any consistent requirement for systemic immune-modulant Rx (e.g. systemic steroids, phototherapy, Cyclosporine)
* History of use of biologic therapy (including intravenous immunoglobulin)
* Recent or anticipated concomitant use of systemic therapies that might alter the course of AD
* Recent or current participation in another research study
* Females who are breastfeeding, pregnant, or with plans to get pregnant during the participation in the study
* Subjects with a history of keloid formation
* History of lidocaine, epinephrine or Novocain allergy
* History of allergy to tape or other adhesive materials
* Hand eczema only (no body involvement).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna De Benedetto, Principal Investigator — UF COM Department of Dermatology
Locations (2):
- United States (2):
  - UF HealthStreet, Gainesville, Florida
  - UF Health Springhill, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 were consented but 15 assigned to receive the intervention
Groups:
- Topical Administration of Study Drug: 2.5 grams of Nanodox 1% (doxycycline monohydrate hydrogel) will be applied topically to an indicated lesion daily for 28 days
  Nanodox 1% (doxycycline monohydrate hydrogel): Subjects will be asked to apply NanoDOX® Hydrogel 1% daily for up to four weeks or until complete clearance whichever is sooner
Period: Overall Study
Arm/Group | Topical Administration of Study Drug
Started | 15
Completed | 13
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: 23 pts signed consent. 8 did not qualify. 2 withdrew from the study before completion. Results are based on 15 subjects
Arm/Group | Topical Administration of Study Drug
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/ Alaskan Native | 0
  Asian | 3
  Native Hawaiian or OPI | 0
  Black or African American | 3
  White | 15
  More than one Race | 1
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 23
Baseline Investigator's Global Assessment "IGA" for Target Area [Count of Participants; unit: Participants]
  Clear | 5
  Almost Clear | 1
  Mild | 9
  Moderate | 5
  Severe | 1
  Not performed | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Description: comparing dermatological scores of treated lesions vs non treated lesions and treated peri-lesional areas with non-treated non-lesional areas
Time Frame: up to 4 weeks of study drug use
Population: 0 pts with treatment related adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Administration of Study Drug
Number analyzed (Participants) | 15
Participants | 0

2. Secondary Outcome: Number of Participants With Reduction in Growth of Skin Flora Including S.Aureus
Description: (positive or negative), difference in number of growth (0 to 3+++)
Time Frame: up to 4 weeks of study drug use
Population: Number of patients with reduction in growth of skin flora including S.Aureus
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects Received Active Drug: Topical Treatment with NanoDox for 14 to 28 days
Arm/Group | All Subjects Received Active Drug
Number analyzed (Participants) | 15
Participants
  Reduction of Staph species | 7
  Reduction of Other flora | 2
  No growth or normal flora at V1 | 6

3. Secondary Outcome: Number of Participant With a Change in Investigator's Global Assessment (IGA) in Target Area
Description: 1 point reduction of IGA score in Target area pre-treatment compared to post treatment (v3)
Time Frame: 4 weeks of topical therapy
Measure: Count of Participants; unit: Participants
Groups:
- All Subjects Received Active Drug: Treated with Nanodox topical for 14 to 28 days
Arm/Group | All Subjects Received Active Drug
Number analyzed (Participants) | 15
Participants
  Reduction of 1 pt | 6
  Reduction of </=2 pt | 7
  no reduction in IGA | 1
  Worsening of IGA | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over 18 months encompassing all 15 included patients receiving drug
Description: 2 subjects were withdrawn early for adverse event "eczema flare-requiring steroid systemic treatment". Other adverse events include upper respiratory infection (2 subjects) requiring treatment. All adverse events considered unlikely/ not related to study drug.
Arm/Group | Topical Administration of Study Drug
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Administration of Study Drug (N=15)
eczema flare-requiring steroid systemic treatment (Skin and subcutaneous tissue disorders) | 2 (2)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/11/NCT02910011/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-11-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT02910011/Prot_SAP_001.pdf